CLINICAL TRIAL: NCT03623256
Title: Comparison of Intrathecal Versus Epidural Fentanyl: Effect of Neuraxial Route of Administration on Fetal Bradycardia in Labor Combined Spinal Epidural Analgesia
Brief Title: Comparison of Intrathecal Versus Epidural Fentanyl on Fetal Bradycardia in Labor Combined Spinal Epidural Analgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor Department of Anesthesiology and Perioperative Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1238162
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Labor Pain; Obstetric Pain
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of four groups:
  Group A: Spinal dose of preservative-free fentanyl 25 mcg. Group B: Spinal preservative-free 0.25% bupivacaine. Group C: Spinal combination of preservative-free 0.25% bupivacaine and fentanyl 25 mcg.
  Group D: Spinal preservative-free 0.25% bupivacaine and epidural fentanyl 100 mcg.
  After the procedure, we will monitor the fetal heart rate and tocometry tracings for 30 min. Thereafter, an epidural infusion with a solution containing 0.125% bupivacaine and 2mcg/mL of fentanyl will be started. We will record demographic variables (age, and BMI), obstetric variables (parity, gestational age, cervical dilation, oxytocin infusion) and anesthetic variables (level of insertion of epidural catheter). We will also record level of insertion, blood pressure every 5 minutes, dermatomal level, pain level, patient satisfaction level and pruritus.
Who Masked: Participant
Masking Description: Participant will be blinded. The investigators will not be blinded because they are the same care providers. In addition, the volume of intrathecal anesthetic is different when bupivacaine plus fentanyl is used in comparison with only one medication used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Spinal Fentanyl (Active Comparator): Spinal dose of preservative-free fentanyl 25 mcg (Volume 0.5 mL)
  Interventions: Drug: Spinal fentanyl
- Spinal Bupivacaine (Active Comparator): Spinal dose of preservative-free 0.25% bupivacaine (Volume 0.5 mL)
  Interventions: Drug: Spinal bupivacaine
- Spinal Fentanyl and Bupivacaine (Active Comparator): Spinal combination of preservative-free 0.25% bupivacaine (0.5 mL) and fentanyl 25 mcg (0.5 mL). (Total Volume 1 mL).
  Interventions: Drug: Spinal Fentanyl and Bupivacaine
- Epidural fentanyl /spinal bupivacaine (Experimental): Spinal preservative-free 0.25% bupivacaine (Volume 0.5 mL) and epidural fentanyl 100 mcg (Volume 2 mL).
  Interventions: Drug: Epidural fentanyl /spinal bupivacaine

INTERVENTIONS:
Drug: Spinal fentanyl — 25 mcg of fentanyl (0.5 mL) will be administered by intrathecal route.
  Other Names: Fentora
  Arms: Spinal Fentanyl
Drug: Spinal bupivacaine — 1.25 mg of preservative-free bupivacaine 0.25% (0.5 mL) will be administered by intrathecal route.
  Other Names: Marcaine
  Arms: Spinal Bupivacaine
Drug: Spinal Fentanyl and Bupivacaine — 1.25 mg of preservative-free bupivacaine 0.25% (0.5 mL), and 25 mcg of fentanyl (0.5 mL) will be administered by intrathecal route.
  Other Names: Marcaine and Fentora
  Arms: Spinal Fentanyl and Bupivacaine
Drug: Epidural fentanyl /spinal bupivacaine — 1.25 mg of preservative-free bupivacaine 0.25% (0.5 mL) will be administered by intrathecal route, and 100 mcg of fentanyl (2 mL) will be administered by epidural route.
  Other Names: Marcaine and Fentora
  Arms: Epidural fentanyl /spinal bupivacaine

SUMMARY:
There have been studies reporting that combined spinal-epidural (CSE) with fentanyl and bupivacaine produce fetal bradycardia, (M.Kuczkowski, 2004) (Abrão K, 2009 ). It is unknown whether any differences in risk exist between fentanyl and bupivacaine when used as a part of the CSE procedure. Some authors have reported cases of parturients who developed uterine hyperactivity and fetal bradycardia after subarachnoid administration of fentanyl during labor. (D'Angelo & Eisenach, 1997) (Friedlander JD, 1997). It has been suggested that uterine hypertonus, leading to non-reassuring fetal heart rate tracings, might be an etiologic factor in these situations. (Landau, 2002).

We propose this study to test the hypothesis that administration of epidural fentanyl is associated with a lower incidence of fetal bradycardia compared to intrathecal fentanyl.

DETAILED DESCRIPTION:
After approval by the Institutional Review Board and written informed consent, we plan to prospectively study pregnant patients who undergo neuraxial labor analgesia. All patients will receive combined-spinal-epidural analgesia. Patients will be randomly assigned to one of four groups by means of sealed envelope technique. Group A will receive a spinal dose of preservative-free fentanyl 25 mcg. Group B will receive one dose of spinal preservative-free 0.25% bupivacaine. Group C will receive a spinal combination of preservative-free 0.25% bupivacaine and fentanyl 25 mcg. Group D will receive spinal preservative-free 0.25% bupivacaine and epidural fentanyl 100 mcg. After the procedure, we will monitor the fetal heart rate and tocometry tracings for 20 min. Thereafter, an epidural infusion with a solution containing 0.125% bupivacaine and 2mcg/mL of fentanyl will be started. We will record demographic variables (age, and BMI), obstetric variables (parity, gestational age, cervical dilation, oxytocin infusion) and anesthetic variables (level of insertion of epidural catheter).

Primary outcomes:

Fetal heart rate (baseline, minimal and abnormal patterns)

Secondary outcomes:

* Blood pressure (systolic, diastolic and mean) measured at baseline and every 5 minutes after administration of medication.
* Dermatomal level measured after 20 minutes of medication administration.
* Pain level (visual analogue scale) after 20 minutes of medication administration.
* Patient satisfaction level (1-10 scale) after 20 minutes of medication administration.
* Uterine tone measured with tocometer at baseline and during 20 minutes after medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Term pregnancy (> 37 weeks)
* Absence of obstetric morbidities
* Active labor
* Request of neuraxial analgesia per patient and/or obstetrician
* Combined spinal-epidural technique

Exclusion Criteria:

* Abnormal fetal heart rate tracing.
* Uterine tachysystole before neuraxial analgesia.
* Baseline blood pressure <90/60 mmHg.
* Allergies to local anesthetics or fentanyl.
* Maternal fever.
* Pruritus before performance of neuraxial analgesia.
* Contraindications for neuraxial technique.
* Unwillingness to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients in labor
Enrollment: 558 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Fetal heart rate | 20 minutes (Starting from placement of labor neuraxial block)
  Fetal bradycardia and abnormal fetal heart rate tracing

SECONDARY OUTCOMES:
Blood pressure | 20 minutes (Starting from placement of labor neuraxial block)
  Maternal systolic, diastolic and mean arterial pressure measured at baseline and every 5 minutes after administration of medication
Dermatomal level | 20 minutes (Starting from placement of labor neuraxial block)
  Analgesic level measured by sensitivity to temperature stimulus
Maternal Pain level: visual analogue scale | 20 minutes (Starting from placement of labor neuraxial block)
  Pain evaluated by visual analogue scale (0, no pain; 10, worst pain)
Patient satisfaction level: Likert Scale | 20 minutes (Starting from placement of labor neuraxial block)
  Satisfaction level measured by Likert Scale (5: fully satisfied, 4: satisfied, 3: neutral, 2: dissatisfied, 1: fully dissatisfied)
Uterine tone | 20 minutes (Starting from placement of labor neuraxial block)
  Measured with tocometer (In milimeters above baseline) at baseline and during 20 minutes after medication administration.

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Riveros Perez, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
The study team will decide about sharing information upon request